CLINICAL TRIAL: NCT06079476
Title: An Open-label, Single-arm, Multicenter Phase 4 Study to Evaluate Safety and Tolerability of Romosozumab (EVENITY® ) in Postmenopausal Women in India With Osteoporosis and a High Risk of Fracture.
Brief Title: A Study of Romosozumab (EVENITY®) in Postmenopausal Women in India With Osteoporosis at a High Risk of Fracture.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210025
Record Dates: First submitted 2023-09-25; First posted 2023-10-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Romosozumab; EVENITY®; Osteoporosis; Women Health
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — romosozumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Phase 4: Romosozumab (Experimental): Participants will be dosed with two subcutaneous (SC) injections of romosozumab once a month for 12 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Single-use prefilled syringe for SC injection.

SUMMARY:
The primary objective of this study is to characterize safety and tolerability of romosozumab in postmenopausal women with osteoporosis and a high risk of fracture in India.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with osteoporosis who are postmenopausal and have a high risk of fracture who provided inform consent (in-person or through their legally authorized representative) to participate in the use of romosozumab per local label in India.

Exclusion Criteria:

* Participants who experienced myocardial infarction or stroke within a year prior to entering this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAE) | Up to 12 months
Number of Participants Experiencing Treatment-emergent Serious Adverse Events (TESAE) | Up to 12 months
Number of Participants Experiencing Clinically Significant Changes in Laboratory Assessments | Baseline, Month 12
Number of Participants With Clinically Significant Changes in Vital Signs | Baseline, Month 12

SECONDARY OUTCOMES:
Percentage Change From Baseline in Bone Mineral Density (BMD) (Measured by Dual-energy X-ray Absorptiometry [DXA]) of the Lumbar Spine | At 6 months and 12 months
Percentage Change From Baseline in BMD (Measured by DXA) of the Total Hip | At 6 months and 12 months
Percentage Change From Baseline in BMD (Measured by DXA) of the Femoral Neck | At 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- India (10):
  - Stavya Spine Hospital and Research Institute SSHRI, Ahmedabad, Gujarat
  - MS Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - King Edward Memorial Hospital And Seth Gordhandas Sunderdas Medical College, Mumbai, Maharashtra
  - Sancheti Institute for Orthopedics and rehabilitation, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Post Graduate Institute of Medical Education and Research, Chandigarh, Punjab
  - MGM Healthcare, Chennai, Tamil Nadu
  - Christain Medical College, Vellore, Tamil Nadu
  - King Georges Medical University, Lucknow, Uttar Pradesh

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com